CLINICAL TRIAL: NCT05442931
Title: Comparison Between Single Dose Pregabalin and Magnesium Sulfate in Controlled Hypotension During Functional Endoscopic Sinus Surgery
Brief Title: Comparison Between Pregabalin and Magnesium Sulfate in Hypotensive Anaesthesia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Eman G Hassan , MD, principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 55:2021
Record Dates: First submitted 2022-03-25; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Functional Endoscopic Sinus Surgery
MeSH Terms: interventions — Pregabalin; Magnesium Sulfate; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Pregabaline (Experimental): Preoperative oral dose of pregabalin for control blood pressure and decrease dose of nitroglycerine consumption
  Interventions: Drug: Pregabalin 150mg
- Magnesium sulfate (Experimental): Preoperative intravenous dose for control blood pressure and heart rate
  Interventions: Drug: Magnesium Sulfate
- Nitroglycrine (Experimental): Measuring the total dose of nitroglycerine used, using a syringe pump
  Interventions: Drug: Nitroglycerin; Other: surgeon satisfaction

INTERVENTIONS:
Drug: Pregabalin 150mg — The oral tablet half an hour preoperative 150 milligrams
  Other Names: Lyrica 150mg
  Arms: Pregabaline
Drug: Magnesium Sulfate — Intravenous administration half an hour preoperative 2 grams
  Other Names: Magnisol 1gm/ 5ml
  Arms: Magnesium sulfate
Drug: Nitroglycerin — measure total dose of nitroglycerine in milligrams using a syringe pump
  Other Names: Nitronal
  Arms: Nitroglycrine
Other: surgeon satisfaction — surgeon satisfaction measured according to Likert's scale
  Other Names: surgeon satisfaction Likert's scale
  Arms: Nitroglycrine

SUMMARY:
Comparison between pregabalin and magnesium sulfate in hypotensive anaethesia

DETAILED DESCRIPTION:
compare the effect of a single-dose 150 mg oral pregabalin and 2 grams intravenous magnesium sulfate given 30 minutes before induction of anesthesia on the total nitroglycerine used in patients undergoing functional endoscopic sinus surgery

ELIGIBILITY:
Inclusion Criteria:

* ASA: class 1 or 2
* Sex: male and female
* Age: from 18 to 70 years
* Patients scheduled for functional endoscopic sinus surgery

Exclusion Criteria:

* Patient on diuretics, corticosteroid, pregabalin
* Patients with a history of allergy to the study drug
* Pregnancy or breastfeeding women Patients with hypertension, cardiac, renal endocrinal diseases
* uncooperative patients (cant does not administer oral tablet)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Dose of nitroglycerine | an hour and half
  total dose measured by a syringe pump

SECONDARY OUTCOMES:
quality of surgical field | an hour and half
  using Boezaart et al grading scale
surgeon satisfaction | an hour and half
  using Likert's scale

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Omar, M.D., Study Director — Minia University
Locations (1):
- Faculty of medicine, Minya, Egypt